CLINICAL TRIAL: NCT03599258
Title: Comparison of Phototherapy Using Neolight Skylife Versus Standardized Phototherapy for Hyperbilirubinemia in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Neolight (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Skylife-2018-001
Record Dates: First submitted 2018-07-11; First posted 2018-07-26 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Jaundice, Neonatal; Neonatal Hyperbilirubinemia; Neonatal Disorder
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal; Infant, Newborn, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm 1 (Other): Skylife device
  Interventions: Device: Skylife
- Arm 2 (Active Comparator): Standard therapy
  Interventions: Device: Standard Therapy

INTERVENTIONS:
Device: Skylife — Newly FDA approved device
  Arms: Arm 1
Device: Standard Therapy — Both devices are considered standard therapy
  Other Names: Natus-Neo Blue Blanket; GE Bili Soft Blanket
  Arms: Arm 2

SUMMARY:
Phototherapy has served as a primary treatment for hyperbilirubinemia in newborn populations. The light emitted through phototherapy interacts with bilirubin at the skin level to transform it into water-soluble products eliminated in urine and stool. Efficacy of phototherapy relies on the irradiance dispensed at the skin level by the treatment and on the surface area of skin exposed. The purpose of this Investigator-initiated, prospective, two-arm, randomized control investigation is to compare the effect of a novel, newly available, FDA cleared, phototherapy device (Neolight Skylife) with the standard phototherapy treatments used in HonorHealth newborn nurseries (Natus-Neo Blue Blanket and GE Bili Soft Blanket) on healthy, newborns ≥ 35 weeks + 0 days Gestational Age (GA) at the time of birth in the treatment of hyperbilirubinemia. We hypothesize that the unconjugated bilirubin level will be comparably reduced across each treatment arm from baseline to 12 and 24 hour intervals.

DETAILED DESCRIPTION:
This is an investigator-initiated, prospective, two-arm randomized control investigation to examine the mean values in patients' unconjugated bilirubin level for a new, FDA cleared device (Neolight Skylife) with the standard phototherapy treatment. Patient data on unconjugated bilirubin level, pressure ulcer and body temperature will be evaluated at baseline, 12-hours post-intervention, 24 hours post-intervention and at discharge.

Neolight Skylife is a compact device that offers phototherapy to infants across all neonatal beds, supplanting multiple, enclosure specific phototherapy devices. Neolight Skylife weighs less than 10 lbs. and is ergonomically designed for portability that allows for easy carrying of the device between beds. Neolight Skylife offers the choice between treatment intensity levels. Neolight Skylife utilizes blue Light-Emitting Diodes (LEDs) to achieve low irradiance of 30 plus or minus 5 μw/cm²/nm, and high irradiance of 45 plus or minus 10, μw/cm²/nm. Neolight Skylife emits light in a narrow bandwidth between 430-475 nm. This light bandwidth corresponds to the spectral absorption of light by bilirubin, and is thus considered to be the most effective for treatment. Neolight Skylife eliminates the risk of UV exposure typically seen with phototherapy treatment through the use of blue LEDs, as this light source does not emit significant energy in the ultraviolet (UV) spectrum. However, as with all phototherapy treatment, protective eye coverings are used to protect the baby's eyes from excessive light exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of at least one parent/legal guardian's signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Infants born after 35 weeks and 0 days of gestation
4. Infants who developed significant hyperbilirubinemia Infants who developed significant hyperbilirubinemia per BiliToolTM plot requiring phototherapy as determined by the attending neonatologist utilizing the American Academy of Pediatrics'

   1. Management of Hyperbilirubinemia in the Newborn Infant 35 or More Weeks of Gestation (Bhutani Nomogram)
   2. Guidelines for Phototherapy in Hospitalized Infants of 35 or More Weeks Gestation

Exclusion Criteria:

Participants will be screened on the following exclusion criteria at the time of enrollment:

* Perinatal asphyxia (Apgar score <4 at 1 minute or <7 at 5 minutes)
* Respiratory distress
* Exchange transfusion
* Major congenital malformations

As identified throughout the course of the investigation, additional exclusion criteria include:

* Direct-reacting component of bilirubin >2 mg/dL
* Glucose-6-phosphate deficiency
* ABO incompatibility
* Evidence of hemolysis
* Evidence of sepsis
* Rhesus hemolytic disease
* Pyruvate kinase deficiency
* Severe dehydration

Ages: 0 Minutes to 7 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Change in unconjugated bilirubin level from pre-test to post-test | Assessment of the endpoint will occur at baseline, 12 hours following treatment, and 24 hours following initial treatment or prior to discharge.
  heel stick blood draw for unconjugated bilirubin level

SECONDARY OUTCOMES:
Maintain body temperature between 97.3F and 99.3F | Assessment of the endpoint will occur at baseline, 12 hours following treatment, and 24 hours following initial treatment or prior to discharge.
  monitor body temperature using a temperature monitoring device
Absence of skin irritation or ulceration | Assessment of the endpoint will occur at baseline, 12 hours following treatment, and 24 hours following initial treatment or prior to discharge.
  visual assessment of the skin for changes

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Abrams, MD, Principal Investigator — Affiliated Physician
Locations (2):
- United States (2):
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - HonorHealth Scottsdale Shea Medical Center, Scottsdale, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abrams M, Gosselin K, Roth CK, Hoffman N. A Randomized Trial Comparing NeoLight Skylife and Blanket Phototherapy in Newborn Indirect Hyperbilirubinemia. Clin Pediatr (Phila). 2024 Jun;63(6):774-778. doi: 10.1177/00099228231190120. Epub 2023 Jul 31. PMID 37522330